CLINICAL TRIAL: NCT06069596
Title: Evaluation of the Effectiveness of Obstetric Lubricant Gel in Labor in Nulliparous and Primiparous Women: A Randomized Controlled Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, kaan baydemir, Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 290819912
Record Dates: First submitted 2023-09-28; First posted 2023-10-06 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Parturition; Obstetric; Injury Pelvic Floor
Keywords: birth; parturition; obstetric lubricant gel; duration of second stage of labor; labor

STUDY DESIGN:
Intervention Model Description: The participants were divided into two groups based on their parity; nulliparous and primiparous. At the outset, each group had 110 participants. Nulliparous and primiparous groups were randomly assigned to two groups as study and control groups by using a computer generating random number table. Obstetric lubricant gel was applied to patients in the study groups. Perinatal outcomes and durations of the labor were compared between study and control groups.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization was performed using a computer program. Accordingly, the study group patients were administered Obstetric gel. The researcher administering Obstetric gel ensured the blinding of healthcare providers and other researchers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): obstetric lubricant gel was applied to patients in the study groups, which had 47 nulliparous and 50 primiparous patients.
  Interventions: Combination Product: Natalis Obstetric Lubrican Gel
- Control group (No Intervention): obstetric lubricant gel was not applied to patients in the control groups, which had 55 nulliparous and 43 primiparous patients.

INTERVENTIONS:
Combination Product: Natalis Obstetric Lubrican Gel — The obstetric lubricant gel was applied to the vaginal canal with a special applicator at the beginning of the active phase of the labor. The gel used in the study was highly viscose and isotonic with a slight acid pH of 6.0 - 6.7 and contained hydroxyethylcellulose, propylene glycol, glycerin. The gel box contained a sterile syringe (15 ml) and a flexible applicator.
  Arms: Study group

SUMMARY:
The investigators hypothesized that the application of lubricant gels at the beginning of the active phase of the labor may reduce duration of the delivery and episiotomy rates. The aim of this study is to investigate and confirm this hypothesis through a randomised controlled trial.

All participants in the study received standard routine antepartum care in the delivery room. Obstetric lubricant gel was applied to patients in the study groups, which had 47 nulliparous and 50 primiparous patients. Perinatal outcomes were compared between the groups.

DETAILED DESCRIPTION:
The participants were divided into two groups based on their parity: nulliparous and primiparous. Initially, each group had 110 participants. Nulliparous and primiparous groups were randomly assigned to two groups as study and control groups using a computer-generated random number table. In this randomized controlled trial, participant allocation was carried out using a computer program to ensure a randomized and unbiased selection process. The randomization procedure was conducted in a double-blind manner, with the study investigators remaining unaware of the allocation until the conclusion of the study. All participants in the study received standard routine antepartum care in the delivery room. Among all patients, 25 participants were lost to follow-up during the study. Consequently, obstetric lubricant gel was applied to patients in the study groups, which included 47 nulliparous and 50 primiparous patients. Perinatal outcomes were compared between the groups

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous and primiparous singleton pregnancies between 37 and 41 weeks + six days of gestation and vertex presentation of fetus with an estimated birth weight of 2000 - 4500g were included in the study

Exclusion Criteria:

* Multiparous pregnancies and women who had ceserean section before and/or contraindication for vaginal delivery were excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
The duration of the active phase of the first stage of labor was compared between the study and control groups | 0 to 600 minutes
  The active phase of labor begins when the cervical dilation is between 4-6 cm and refers to the time elapsed until full cervical dilation.
The duration of the second stage of labor was compared between the study and control groups | 0 to 240 minutes
  The second stage of labor begins when the cervical dilation is complete and continues until the birth of the newborn.

SECONDARY OUTCOMES:
Episiotomy rates | Episiotomy is a technique performed during the second stage of labor.
  differences between study and control groups

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seval MM, Yuce T, Yakistiran B, Sukur YE, Ozmen B, Atabekoglu C, Koc A, Soylemez F. Effects of obstetric gel on the process and duration of labour in pregnant women: Randomised controlled trial. J Obstet Gynaecol. 2017 Aug;37(6):714-718. doi: 10.1080/01443615.2017.1288711. Epub 2017 Mar 21. PMID 28325124
- [Background] Azarkish F, Janghorban R, Bozorgzadeh S, Merbalouchzai F, Razavi M, Badiee M. Effect of lubricant gel on the length of the first stage of labour and perineal trauma in primiparous women. J Obstet Gynaecol. 2022 Jul;42(5):867-871. doi: 10.1080/01443615.2021.1946021. Epub 2021 Sep 27. PMID 34569413